CLINICAL TRIAL: NCT03916601
Title: A Randomized, Double-blind, Single-dose, Cross-over Study in Two Cohorts to Compare Exposure and Activity of SAR341402 Mix 70/30 to Novolog® Mix 70/30, Novomix® 30 and SAR341402 Rapid-Acting Solution Using the Euglycemic Clamp Technique, in Patients With Type 1 Diabetes Mellitus
Brief Title: Comparison of Exposure and Activity of SAR341402 Mix 70/30 to NovoLog Mix 70/30, NovoMix 30 and SAR341402 Rapid-acting Solution in Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PDY15084; 2017-002482-22; U1111-1197-7984 (Other: UTN)
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart; insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Test (T) (Experimental): SAR341402 Mix 70/30: single dose injection
  Interventions: Drug: SAR341402
- Reference 1 (R1) (Active Comparator): NovoLog Mix 70/30: single dose injection
  Interventions: Drug: Insulin Aspart
- Reference 2 (R2) (Active Comparator): NovoMix30: single dose injection
  Interventions: Drug: Insulin Aspart
- Reference 3 (R3) (Experimental): SAR341402 rapid-acting solution: single dose injection
  Interventions: Drug: SAR341402

INTERVENTIONS:
Drug: SAR341402 — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
  Arms: Reference 3 (R3)
Drug: Insulin Aspart — Pharmaceutical form: suspension for injection
  Route of administration: subcutaneous
  Other Names: NovoLog Mix 70/30
  Arms: Reference 1 (R1)
Drug: Insulin Aspart — Pharmaceutical form: suspension for injection
  Route of administration: subcutaneous
  Other Names: Novo Mix 30
  Arms: Reference 2 (R2)
Drug: SAR341402 — Pharmaceutical form: suspension for injection
  Route of administration: subcutaneous
  Arms: Test (T)

SUMMARY:
Primary Objectives:

* To demonstrate similarity in exposure of SAR341402 Mix 70/30 to NovoLog Mix 70/30 and NovoMix 30 (cohort 1).
* To demonstrate distinctiveness in early and intermediate exposure of SAR341402 Mix 70/30 compared to SAR341402 rapid-acting solution (cohort 2).

Secondary Objectives:

* To demonstrate similarity in activity of SAR341402 Mix 70/30 to NovoLog Mix 70/30 and NovoMix 30.
* To demonstrate distinctiveness in early and intermediate activity of SAR341402 Mix 70/30 compared to SAR341402 rapid-acting solution.
* To assess the safety and tolerability of SAR341402 rapid-acting solution and SAR341402 Mix 70/30.

DETAILED DESCRIPTION:
* Cohort 1: The total study duration for a screened patient will be about 3 - 8 weeks (excluding screening), with screening period of 4 to 28 days, 3 treatment periods of 2 days each period, washout period of 5 to 18 days, and end-of-study visit at 5 to 12 days after last IMP administration.
* Cohort 2: The total study duration for a screened patient will be about 2 - 5 weeks (excluding screening), with screening period of 4 to 28 days, 2 treatment periods of 2 days each period, washout period of 5 to 18 days, and end-of-study visit at 5 to 12 days after last IMP administration.

ELIGIBILITY:
Inclusion criteria :

* Total insulin dose of < 1.0 U/kg/day.
* Total basal insulin dose ≤0.4 U/kg/day.
* Fasting serum C-peptide < 0.3 nmol/L.
* Anti-insulin antibody titer ≤30.0 kU/L.
* Glycohemoglobin (HbA1c) ≤ 9%.
* Stable insulin regimen for at least 2 months prior to study.
* Normal findings in medical history and physical examination (cardiovascular system, chest and lungs, thyroid, abdomen, nervous system, skin and mucosae, and musculo-skeletal system), vital signs, electrocardiogram (ECG) and safety lab.

Exclusion criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic (apart from diabetes mellitus type 1), hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, or infectious disease, or signs of acute illness.
* More than one episode of severe hypoglycemia with seizure, coma or requiring assistance of another person during the past 6 months and/or hospitalized for diabetic ketoacidosis.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month).
* Symptomatic postural hypotension, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥30 mmHg within 3 minutes when changing from supine to standing position.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.
* Likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol.
* Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication, with the exception of insulins, thyroid hormones, lipid-lowering and antihypertensive drugs and if female with the exception of hormonal contraception or menopausal hormone replacement therapy.
* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
(Cohort 1) Assessment of PK parameter: Maximum insulin concentration (INS-Cmax) | 24 hours
  Maximum plasma concentration (Cmax) of SAR341402 Mix 70/30, NovoLog Mix 70/30, NovoMix 30 and SAR341402 within 24 hours
(Cohort 1) Assessment of PK parameter: Area under the insulin concentration time curve (INS-AUClast) | 0 to 24 hours
  INS-AUC of SAR341402 Mix 70/30, NovoLog Mix 70/30, and NovoMix 30 from 0 to 24 hours
(Cohort 2) Assessment of PK parameters: Area under the insulin concentration time curve from 0 to 4 hours post administration (INS-AUC0-4H) | 0 to 4 hours
  INS-AUC0-4H for SAR341402 Mix 70/30 and SAR341402 rapid acting solution from 0 to 4 hours
(Cohort 2) Area under the insulin concentration time curve from 4 to 12 hours post administration (INS-AUC4-12H) | 4 to 12 hours
  INS-AUC4-12H for SAR341402 Mix 70/30 and SAR341402 rapid acting solution from 4 to 12 hours
(Cohort 2) Assessment of PK parameter: Maximum insulin concentration (INS-Cmax) | 24 hours
  (Cohort 2) Maximum plasma concentration (Cmax) of SAR341402 Mix 70/30 and SAR341402 rapid acting solution within 24 hours

SECONDARY OUTCOMES:
Assessment of PK parameter: Area under the insulin concentration time curve from 0 to infinity (INS-AUC) | 0 to 24 hours
  (Cohort 1) INS-AUC for SAR341402 Mix 70/30, Novolog Mix 70/30 and NovoMix 30 from 0 to 24 hours
Assessment of PK parameter: Area under the insulin concentration time curve for fractional periods post administration (INS-AUC0-4H, INS-AUC0-24H, INS-AUC4-24H) | 0 to 4 hours, 0 to 24 hours, and 4 to 24 hours
  (Cohort 1) INS-AUC0-4H, INS-AUC0-24H, INS-AUC4-24H for SAR341402 Mix 70/30, Novolog Mix 70/30 and NovoMix 30
Assessment of PK parameter: Time to INS-Cmax | 24 hours - 4. 24 hours - 5. 0 to 24 hours - 6. 24 hours - 7. 24 hours - 8. 24 hours - 9. 0 to 4 hours - 10. 4 to 12 hours - 11. 24 hours - 12. 24 hours -
  (Cohort 1) INS-tmax for SAR341402 Mix 70/30, Novolog Mix 70/30, NovoMix 30 and SAR341402 rapid acting solution within 24 hours
Assessment of PK parameter: Half-life (t1/2) | 24 hours
  (Cohort 1) INS-t1/2z for SAR341402 Mix 70/30, Novolog Mix 70/30 and NovoMix 30 within 24 hours
Assessment of PD parameter: GIR versus time curve from 0 to 24 hours post administration (GIR-AUC0-24H) | 0 to 24 hours
  (Cohort 1) The area under the body weight standardized glucose infusion rate (GIR) versus time curve from 0 to 24 hours post administration for SAR341402 Mix 70/30, Novolog Mix 70/30 and NovoMix 30 from 0 to 24 hours
Assessment of PD parameter: Maximum smoothed body weight standardized glucose infusion rate (GIRmax) | 24 hours
  (Cohort 1) GIRmax for SAR341402 Mix 70/30, Novolog Mix 70/30, NovoMix 30 and SAR341402 rapid acting solution within 24 hours
Assessment of PD parameter: Time to GIRmax (GIR-tmax) | 24 hours
  (Cohort 1) GIR-tmax for SAR341402 Mix 70/30, Novolog Mix 70/30, NovoMix 30 and SAR341402 rapid acting solution within 24 hours
Assessment of PK parameter: Time to Cmax (INS-tmax) | 24 hours
  (Cohort 2) INS-tmax for SAR341402 Mix 70/30 and SAR341402 rapid acting solution within 24 hours
Assessment of PD parameter: The area under the body weight standardized glucose infusion rate (GIR) versus time curve from 0 to 4 hours post administration (GIR-AUC0-4H) | 0 to 4 hours
  (Cohort 2) GIR-AUC0-4H for SAR341402 Mix 70/30 and SAR341402 rapid acting solution from 0 to 4 hours
Assessment of PD parameter: The area under the body weight standardized glucose infusion rate (GIR) versus time curve from 4 to 12 hours post administration (GIR-AUC4-12H) | 4 to 12 hours
  (Cohort 2) GIR-AUC4-12H for SAR341402 Mix 70/30 and SAR341402 rapid acting solution from 4 to 12 hours
Assessment of PD parameter: Maximum smoothed body weight standardized glucose infusion rate (GIRmax) | 24 hours
  (Cohort 2) GIRmax for SAR341402 Mix 70/30, Novolog Mix 70/30, NovoMix 30 and SAR341402 rapid acting solution within 24 hours
Assessment of PD parameter: Time to GIRmax (GIR-tmax) | 24 hours
  (Cohort 2) GIR-tmax for SAR341402 Mix 70/30, Novolog Mix 70/30, NovoMix 30 and SAR341402 rapid acting solution within 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 2760001, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Kapitza C, Nosek L, Schmider W, Teichert L, Mukherjee B, Nowotny I. A single-dose euglycaemic clamp study in two cohorts to compare the exposure of SAR341402 (insulin aspart) Mix 70/30 with US- and European-approved versions of insulin aspart Mix 70/30 and SAR341402 rapid-acting solution in subjects with type 1 diabetes. Diabetes Obes Metab. 2021 Mar;23(3):674-681. doi: 10.1111/dom.14260. Epub 2020 Dec 10. PMID 33236518